CLINICAL TRIAL: NCT07117942
Title: The Efficacy and Safety of Different Doses of Fermented Deglycyrrhizinated Licorice (FDGL) in the Management of Diabetic Neuropathy: A Randomized Controlled Trial
Brief Title: FDGL Dose-Finding Study for Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud I Mostafa, Lecturer of Clinical Pharmacy, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6016
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Neuropathy
Keywords: FDGL; Diabetic neuropathy; Pain; Dose-finding
MeSH Terms: conditions — Diabetic Neuropathies; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Matching placebo capsules administered daily for 3 months
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice (FDGL)
- FDGL 400 mg (Experimental): Fermented Deglycyrrhizinated Licorice 400mg daily for 3 months
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice (FDGL)
- FDGL 800 mg (Experimental): Fermented Deglycyrrhizinated Licorice 800mg daily for 3 months
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice (FDGL)
- FDGL 1000 mg (Experimental): Fermented Deglycyrrhizinated Licorice 1000mg daily for 3 months
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice (FDGL)
- FDGL 1200 mg (Experimental): Fermented Deglycyrrhizinated Licorice 1200mg daily for 3 months
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice (FDGL)

INTERVENTIONS:
Drug: Fermented Deglycyrrhizinated Licorice (FDGL) — Fermented Deglycyrrhizinated Licorice (FDGL) in oral powder capsules; prepared through three consecutive steps: fermentation of licorice roots, removal of glycyrrhizinic acid content (deglycyrrhizination), and lyophilization according to EUROPEAN PATENT SPECIFICATION Ep 1 925 312 B

SUMMARY:
This study investigates the optimal dose of fermented deglycyrrhizinated licorice (FDGL) that maximizes both safety and efficacy in managing diabetic neuropathy complications in adults. The study is a single-center, double-blind, parallel, placebo-controlled randomized clinical trial where patients with diabetic neuropathy are randomized to receive placebo, 400 mg, 800 mg, 1000 mg, or 1200 mg daily doses of FDGL for three months. The primary objective is to determine the percentage improvement of diabetic neuropathy presentations and pain scores at three months relative to baseline.

DETAILED DESCRIPTION:
This is a single-center, double-blinded, parallel, randomized clinical trial conducted at Al-Hussein University Hospital, Cairo, Egypt. Eligible patients are randomized to receive either placebo, 400 mg, 800 mg, 1000 mg, or 1200 mg daily FDGL doses in a 1:1:1:1:1 ratio using block randomization with a block size of 5. The study employs computer-assisted random number generation for treatment allocation. Both patients and nurses are blinded to treatment allocation, with assignments kept in sealed envelopes opened only at enrollment. The study duration is 3 months with follow-up assessments at 1, 2, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 70 years
* Documented history of type I or type II diabetes mellitus
* Confirmed diagnosis of at least one diabetes-related complication, including peripheral neuropathy
* Diagnosis of peripheral neuropathy confirmed in both lower extremities
* Numeric rating scores (VAS) on 0 to 10 scale ≥ 4 for at least 6 months in feet/legs
* Ability to provide written informed consent
* If using concurrent therapies for diabetic neuropathy (pregabalin, gabapentin, or duloxetine), must be on stable doses for at least 3 months prior to study start

Exclusion Criteria:

* Concomitant chronic kidney disease
* Hepatic impairment
* Heart failure
* Cancer
* Major psychiatric disorders
* Pregnancy
* Refusal to sign informed consent
* Use of non-pharmacologic management strategies for diabetic neuropathy including:

  * TENS (Transcutaneous Electrical Nerve Stimulation)
  * Nerve block procedures
  * Acupuncture
  * Laser therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 1 month, 2 months, and 3 months
  The percentage improvement of diabetic neuropathy symptoms and pain scores (measured on a 0-10 scale where 0 = no pain and 10 = severe pain) at 3 months relative to baseline. This includes assessment of neuropathic complications in both lower extremities.

SECONDARY OUTCOMES:
Incidence of adverse effects | Throughout the 3-month study period
  Percentage of participants experiencing adverse effects including headache, abdominal pain, nausea, or vomiting during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aly Massoud, PhD, Study Chair — Department of Hepato-gastroenterology and Infectious Diseases, Faculty of Medicine, Al-Azhar University, Cairo, Egypt
Locations (1):
- Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Massoud A, Ebiary FHE, Raafat M, et al. The Effect of Fermented Deglycyrrhizinized Liquorice Extract on the Structure of Gastrocnemius Muscle and Sciatic Nerve in Experimentally Induced Diabetes Mellitus in Rats: Histopathological Study. J Cytol Histol 2019;10:1-8.